CLINICAL TRIAL: NCT05361967
Title: Tack Optimized Balloon Angioplasty Post-Market Study
Acronym: TOBA PMS
Status: Terminated | Type: Observational
Why Stopped: Terminated due to slow enrollment
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IGT-00295
Record Dates: First submitted 2022-04-25; First posted 2022-05-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-02

CONDITIONS: PAD - Peripheral Arterial Disease; PAD; Dissection; Arterial Dissection; Peripheral Arterial Disease; Peripheral Vascular Diseases
MeSH Terms: conditions — Dissection, Blood Vessel; Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ATK: Above-The-Knee: Subjects with claudication (Rutherford 3) or CLTI (Rutherford 4 or 5), who have undergone an endovascular procedure utilizing adjunctive therapies, other than balloon angioplasty alone, which are then followed by PTA and IVUS, and have an arterial dissection requiring repair. ATK subjects will have baseline lesions in the superficial femoral and/or proximal popliteal arteries.
  Interventions: Device: The Tack Endovascular System
- BTK: Below-The-Knee: Subjects with CLTI (Rutherford 4 or 5), who have undergone an endovascular procedure utilizing adjunctive therapies, other than balloon angioplasty alone, which are then followed by PTA and IVUS, and have an arterial dissection requiring repair. BTK subjects will have baseline lesions in the mid/distal popliteal, peroneal and/or tibial arteries.
  Interventions: Device: The Tack Endovascular System

INTERVENTIONS:
Device: The Tack Endovascular System — The Tack Endovascular System is designed to treat vascular dissections with Tack implant(s) following angioplasty.

SUMMARY:
The objective of this study is to obtain outcomes following dissection repair with the Tack Endovascular System in a broad population of patients undergoing endovascular treatment of lesions within the superficial femoral, popliteal, peroneal, and/or tibial arteries.

DETAILED DESCRIPTION:
The purpose of this post-market study is to obtain outcomes following dissection repair with the Tack Endovascular System in a broad population of patients undergoing endovascular treatment of lesions within the superficial femoral, popliteal, peroneal, and/or tibial arteries.

The Tack Endovascular System has been shown to effectively repair dissection and improve outcomes in clinical studies. Additional data, such as clinical utility of the Tack Endovascular System with the combined use of adjunctive therapies - other than balloon angioplasty alone, is needed.

Patients with claudication or CLI, who meet Rutherford classification 3, 4, or 5 criteria if ATK and Rutherford classification criteria 4 or 5 if BTK, who have undergone an above the knee (ATK) or below the knee (BTK) endovascular procedure utilizing adjunctive therapies other than balloon angioplasty alone which are then followed by PTA and IVUS, and have an arterial dissection requiring repair.

Approximately 100 subjects will be enrolled in up to 10 sites. The enrollment will be capped as follows:

* ATK: 50% of subjects
* BTK: 50% of subjects

After enrollment of planned 100 subjects and interim analysis, the study may enroll up to 200 additional subjects at up to 20 additional sites, with each site limited to 15% of total enrollment.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Age ≥ 18 years
2. Willingness to comply with study follow-up evaluations at the predefined time intervals
3. Signs the written informed consent
4. Meets Rutherford classification criteria:

   1. ATK subjects can be RCC 3, 4 or 5
   2. BTK subjects must be RCC 4 or 5

Angiographic Inclusion Criteria

1. A de novo or restenotic, non-stented target lesion with pre-intervention stenosis or occlusion (by visual estimate)
2. ATK Lesions:

   1. must be in the superficial femoral and/or proximal popliteal (P1) arteries and
   2. have a reference vessel diameter range of 3.5-6.0mm or 4.0-8.0mm.
3. BTK Lesions:

   1. must be in the mid/distal popliteal (P2/P3), peroneal and/or tibial arteries and
   2. have a reference vessel diameter range of 1.5-4.5mm Note: The mid popliteal artery begins at the superior aspect of the patella.

Post-IVUS Inclusion Criteria

1. Presence of an arterial dissection requiring repair per investigator judgement
2. ATK reference vessel diameter range of 3.5-6.0mm or 4.0-8.0mm
3. BTK reference vessel diameter range of 1.5-4.5mm

Exclusion Criteria:

General Exclusion Criteria

1. Subject is known to be breastfeeding, pregnant or planning to become pregnant during the study
2. Anticipated life expectancy < 12 months
3. Known COVID positive test within 14 days and active symptoms
4. Known renal disease that precludes contrast administration
5. Presence of a wound that in the opinion of the investigator cannot be healed with transmetatarsal amputation (TMA)
6. Contraindication to anticoagulation and/or antiplatelet therapy
7. Known allergy to nitinol (nickel and/or titanium)
8. Known allergy to contrast media that cannot be adequately pre-medicated prior to index procedure
9. Previous or planned surgical or interventional procedure within 3 days before or 30 days after the index procedure.

   Note: this excludes successful inflow artery treatment within the same hospitalization or a documented pre-planned minor amputation.
10. Subject has any condition that in the opinion of the investigator precludes the subject from participation

Angiographic Exclusion Criteria

1. Residual diameter stenosis ≥30% (visual estimate) after PTA
2. Aneurysm, acute or sub-acute thrombosis in target lesion
3. Acute vessel occlusion after PTA not attributed to dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with claudication (Rutherford 3) or CLTI (Rutherford 4 or 5), who have undergone an endovascular procedure utilizing adjunctive therapies, other than balloon angioplasty alone, which are then followed by PTA and IVUS, and have an arterial dissection requiring repair. ATK lesions will be in the superficial femoral and/or proximal popliteal arteries; BTK lesions will be in the mid/distal popliteal, peroneal and/or tibial arteries. To be enrolled, subjects must meet all inclusion criteria and not meet any of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Procedure Success | Measured on Day 0 of enrollment, upon completion of the Index Procedure
  Defined as demonstrated target lesion patency (<30% residual diameter stenosis, by visual estimate) without the use of a bail out stent within the target lesion and without the occurrence of MALE + POD upon completion of the index procedure.

SECONDARY OUTCOMES:
Target Lesion Patency - ATK, 6 Months | 6 Months
  Defined as freedom from duplex ultrasound derived binary restenosis (PSVR ≥ 2.5) within the PTA treated segment, without reintervention
Target Lesion Patency - ATK, 12 Months | 12 Months
  Defined as freedom from duplex ultrasound derived binary restenosis (PSVR ≥ 2.5) within the PTA treated segment, without reintervention
Target Lesion Patency - ATK, 24 Months | 24 Months
  Defined as freedom from duplex ultrasound derived binary restenosis (PSVR ≥ 2.5) within the PTA treated segment, without reintervention
Target Lesion Patency - BTK, 6 Months | 6 Months
  Defined as presence of antegrade blood flow using duplex ultrasound within the PTA treated segment, without reintervention.
Target Lesion Patency - BTK, 12 Months | 12 Months
  Defined as presence of antegrade blood flow using duplex ultrasound within the PTA treated segment, without reintervention.
Target Lesion Patency - BTK, 24 Months | 24 Months
  Defined as presence of antegrade blood flow using duplex ultrasound within the PTA treated segment, without reintervention.
Death | 6 months
  All cause death
Death | 12 months
  All cause death
Death | 24 months
  All cause death
Major Adverse Limb Events | 6 months
  Rate of MALE
Major Adverse Limb Events | 12 months
  Rate of MALE
Major Adverse Limb Events | 24 months
  Rate of MALE
Freedom from clinically driven target lesion revascularization (CD-TLR) - ATK, 6 Months | 6 months
  TLR is defined as re-treatment by an invasive procedure, including atherectomy, angioplasty, intravascular lithotripsy, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen of the target vessel. TLR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as PSVR ≥ 2.5 by DUS or if angiography shows >50% diameter stenosis and there are symptoms attributable to increased ischemia or worsening of ABI (defined as deterioration by more than 0.15 from the maximum post-procedural level) that is clearly referable to the target lesion.
Freedom from clinically driven target lesion revascularization (CD-TLR) - BTK, 6 Months | 6 months
  TLR is defined as re-treatment by an invasive procedure, including atherectomy, angioplasty, intravascular lithotripsy, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen of the target vessel. TLR will be classified as clinically driven or non-clinically driven by the investigator.Clinically driven is defined as a restenosis of ≥ 70% in the target vessel with wound persistence, new wounds or reoccurrence of ischemic rest pain.
Freedom from clinically driven target lesion revascularization (CD-TLR) - ATK, 12 Months | 12 months
  TLR is defined as re-treatment by an invasive procedure, including atherectomy, angioplasty, intravascular lithotripsy, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen of the target vessel. TLR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as PSVR ≥ 2.5 by DUS or if angiography shows >50% diameter stenosis and there are symptoms attributable to increased ischemia or worsening of ABI (defined as deterioration by more than 0.15 from the maximum post-procedural level) that is clearly referable to the target lesion.
Freedom from clinically driven target lesion revascularization (CD-TLR) - BTK, 12 Months | 12 months
  TLR is defined as re-treatment by an invasive procedure, including atherectomy, angioplasty, intravascular lithotripsy, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen of the target vessel. TLR will be classified as clinically driven or non-clinically driven by the investigator.Clinically driven is defined as a restenosis of ≥ 70% in the target vessel with wound persistence, new wounds or reoccurrence of ischemic rest pain.
Freedom from clinically driven target lesion revascularization (CD-TLR) - ATK, 24 Months | 24 months
  TLR is defined as re-treatment by an invasive procedure, including atherectomy, angioplasty, intravascular lithotripsy, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen of the target vessel. TLR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as PSVR ≥ 2.5 by DUS or if angiography shows >50% diameter stenosis and there are symptoms attributable to increased ischemia or worsening of ABI (defined as deterioration by more than 0.15 from the maximum post-procedural level) that is clearly referable to the target lesion.
Freedom from clinically driven target lesion revascularization (CD-TLR) - BTK, 24 Months | 24 months
  TLR is defined as re-treatment by an invasive procedure, including atherectomy, angioplasty, intravascular lithotripsy, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen of the target vessel. TLR will be classified as clinically driven or non-clinically driven by the investigator.Clinically driven is defined as a restenosis of ≥ 70% in the target vessel with wound persistence, new wounds or reoccurrence of ischemic rest pain.
Freedom from clinically driven target vessel revascularization (CD-TVR) - ATK, 6 Months | 6 months
  TVR is defined as a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel, exclusive of the target lesion site. TVR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as PSVR ≥ 2.5 by DUS or if angiography shows >50% diameter stenosis and there are symptoms attributable to increased ischemia or worsening of ABI (defined as deterioration by more than 0.15 from the maximum post-procedural level) that is clearly referable to the target vessel.
Freedom from clinically driven target vessel revascularization (CD-TVR) - BTK, 6 Months | 6 months
  TVR is defined as a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel, exclusive of the target lesion site. TVR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as a restenosis of ≥ 70% in the target vessel with wound persistence, new wounds or reoccurrence of ischemic rest pain.
Freedom from clinically driven target vessel revascularization (CD-TVR) - ATK, 12 Months | 12 months
  TVR is defined as a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel, exclusive of the target lesion site. TVR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as PSVR ≥ 2.5 by DUS or if angiography shows >50% diameter stenosis and there are symptoms attributable to increased ischemia or worsening of ABI (defined as deterioration by more than 0.15 from the maximum post-procedural level) that is clearly referable to the target vessel.
Freedom from clinically driven target vessel revascularization (CD-TVR) - BTK, 12 Months | 12 months
  TVR is defined as a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel, exclusive of the target lesion site. TVR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as a restenosis of ≥ 70% in the target vessel with wound persistence, new wounds or reoccurrence of ischemic rest pain.
Freedom from clinically driven target vessel revascularization (CD-TVR) - ATK, 24 Months | 24 months
  TVR is defined as a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel, exclusive of the target lesion site. TVR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as PSVR ≥ 2.5 by DUS or if angiography shows >50% diameter stenosis and there are symptoms attributable to increased ischemia or worsening of ABI (defined as deterioration by more than 0.15 from the maximum post-procedural level) that is clearly referable to the target vessel.
Freedom from clinically driven target vessel revascularization (CD-TVR) - BTK, 24 Months | 24 months
  TVR is defined as a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel, exclusive of the target lesion site. TVR will be classified as clinically driven or non-clinically driven by the investigator. Clinically driven is defined as a restenosis of ≥ 70% in the target vessel with wound persistence, new wounds or reoccurrence of ischemic rest pain.
Target Limb Salvage | 6 months
  Freedom from above-ankle amputation.
Target Limb Salvage | 12 months
  Freedom from above-ankle amputation.
Target Limb Salvage | 24 months
  Freedom from above-ankle amputation.
Minor Amputation | 6 months
  Freedom from target limb unplanned minor amputation
Minor Amputation | 12 months
  Freedom from target limb unplanned minor amputation
Minor Amputation | 24 months
  Freedom from target limb unplanned minor amputation
Rutherford Classification | 6 months
  Changes from baseline in Rutherford classification
Rutherford Classification | 12 months
  Changes from baseline in Rutherford classification
Rutherford Classification | 24 months
  Changes from baseline in Rutherford classification
Ankle and/or Toe Brachial Index | 6 months
  Changes from baseline in target limb Ankle Brachial Index (ABI) and/or Toe Brachial Index (TBI) measurement at post-procedure
Ankle and/or Toe Brachial Index | 12 months
  Changes from baseline in target limb Ankle Brachial Index (ABI) and/or Toe Brachial Index (TBI) measurement at post-procedure
Ankle and/or Toe Brachial Index | 24 months
  Changes from baseline in target limb Ankle Brachial Index (ABI) and/or Toe Brachial Index (TBI) measurement at post-procedure
Wound Status | 6 months
  Changes from baseline in target limb wound status
Wound Status | 12 months
  Changes from baseline in target limb wound status
Quality of Life / EuroQol EQ-5D-5L | 30 Days
  Changes from baseline in EQ-5D-5L questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Quality of Life / EuroQol EQ-5D-5L | 6 months
  Changes from baseline in EQ-5D-5L questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Quality of Life / EuroQol EQ-5D-5L | 12 months
  Changes from baseline in EQ-5D-5L questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Quality of Life / EuroQol EQ-5D-5L | 24 months
  Changes from baseline in EQ-5D-5L questionnaire. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Adverse Events | Measured on Day 0 of enrollment, upon completion of the Index Procedure
  Device related adverse events (AEs) upon completion of the index procedure

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Advanced Heart and Vein Center - Thornton, Thornton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Palm Vascular Center Research, Fort Lauderdale, Florida
  - Munster Medical Research Foundation, Munster, Indiana
  - Advanced Heart and Vascular Institute of Hunterdon, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Ascension St. John Heart and Vascular Center, Bartlesville, Oklahoma
  - The Miriam Hospital, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - North Dallas Research Associates, McKinney, Texas